CLINICAL TRIAL: NCT04986566
Title: Perioperative Telemonitoring to Optimize Cancer Care and Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20717; NCI-2021-03335 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20717 (Other: City of Hope Medical Center); P30CA033572 (NIH); R21NR019866 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-08-03 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Malignant Digestive System Neoplasm
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (telemonitoring) (Experimental): Patients wear a Vivofit 4 daily for 30 days after hospital discharge for steps monitoring, and complete questionnaires over 5-7 minutes about symptoms and quality of life using the Aetonixx app up to 7 days before surgery, before being discharged from the hospital after surgery, and on days 2, 7, 14, 30 after discharge. Patients also complete pulse oximetry, temperature, blood pressure, heart rate, and weight assessment using at-home monitoring devices before surgery, then on days 2, 7, 14, 30 after discharge. Patients assessments are monitored by the surgical team in real-time to identify outcome trends, including onset, worsening/improving measures, and sporadic versus consistent measures.
  Interventions: Other: Best Practice; Behavioral: Health Education; Other: Medical Device Usage and Evaluation; Other: Quality-of-Life Assessment
- Arm II (enhanced usual care) (Active Comparator): Patients wear a Vivofit 4 for daily steps monitoring, and complete questionnaires over 5-7 minutes about symptoms and quality of life using the Aetonixx app up to 7 days before surgery, before being discharged from the hospital after surgery, and on days 2, 7, 14, 30 after discharge. Patients also complete pulse oximetry, temperature, blood pressure, heart rate, and weight assessment using at-home monitoring devices before surgery, then on days 2, 7, 14, 30 after discharge. Patients use standard procedures for reporting problems.
  Interventions: Other: Best Practice; Behavioral: Health Education; Other: Medical Device Usage and Evaluation; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Best Practice — Use standard reporting procedures
  Other Names: standard of care
Behavioral: Health Education — Use Aetonixx app
Other: Medical Device Usage and Evaluation — Wear Vivofit 4
Other: Quality-of-Life Assessment — Complete questionnaires

SUMMARY:
This study aims to see whether an at-home monitoring program that collects health, symptoms, and quality of life data in real-time can be included as part of the care of surgery patients in order to provide better recovery. Patient-generated health data (weight, temperature, oxygen level, heart rate, blood pressure, daily steps, symptoms, quality of life) using at-home monitoring devices (thermometer, a pulse oximeter, a digital scale and a Vivofit 4 watch) and smart device applications are used more and more to measure value and quality in cancer care. However, measuring patient-generated health data is not currently part of standard care following cancer surgery. An at-home monitoring program may improve the care of patients after hospital discharge from surgery and may help reduce complications by identifying issues early.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To conduct a pilot randomized trial of a remote, perioperative telemonitoring intervention to improve patient-centered outcomes, surgical outcomes, and healthcare resource use in English and Spanish-speaking patients scheduled to undergo major abdominal gastrointestinal (GI) cancer surgery.

Ia. Assess the feasibility, retention, and acceptability of the remote perioperative telemonitoring intervention as measured by the percentage of patients who a) agree to participate; b) complete >= 70% of the telemonitoring; and c) report satisfaction with the intervention through structured exit interviews.

Ib. Determine the preliminary efficacy of the remote perioperative telemonitoring intervention on surgical outcomes, healthcare utilization, patient-reported outcomes (PROs), and functional recovery.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (TELEMONITORING): Patients wear a Vivofit 4 daily for 30 days after hospital discharge for steps monitoring, and complete questionnaires over 5-7 minutes about symptoms and quality of life using the Aetonixx application (app) up to 7 days before surgery, before being discharged from the hospital after surgery, and on days 2, 7, 14, 30 after discharge. Patients also complete pulse oximetry, temperature, blood pressure, heart rate, and weight assessment using at-home monitoring devices before surgery, then on days 2, 7, 14, 30 after discharge. Patients assessments are monitored by the surgical team in real-time to identify outcome trends, including onset, worsening/improving measures, and sporadic versus consistent measures.

ARM II (ENHANCED USUAL CARE): Patients wear a Vivofit 4 for daily steps monitoring, and complete questionnaires over 5-7 minutes about symptoms and quality of life using the Aetonixx app up to 7 days before surgery, before being discharged from the hospital after surgery, and on days 2, 7, 14, 30 after discharge. Patients also complete pulse oximetry, temperature, blood pressure, heart rate, and weight assessment using at-home monitoring devices before surgery, then on days 2, 7, 14, 30 after discharge. Patients use standard procedures for reporting problems.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients scheduled to undergo major abdominal surgery for gastrointestinal (GI) malignancies. GI procedures include esophagectomy, gastrectomy, colectomy, abdominoperineal resection/low anterior resection, hepatectomy, pancreatectomy (distal or pancreaticoduodenectomy), and cytoreductive surgery for peritoneal carcinomatosis. We will include patients scheduled for an ostomy (colostomy or diverting ileostomy)
* Age 18 years or older
* Ability to read and understand English or Spanish
* We are targeting patients across all stages of disease
* Age criterion for this study is based on the National Institute of Health (NIH)'s age criteria, which defines an adult as individuals aged 18 years and over. There are no restrictions related to performance status or life expectancy
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2026-02-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Laleh Melstrom, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 188 eligible patients were approached for study participation. Of these, 54 declined for various reasons: not tech-savvy (n = 2), no time/too busy (n = 13), not interested in clinical research (n = 5), feeling overwhelmed (n = 10), other reasons (n = 6), and two or more of the aforementioned reasons (n = 18). Ultimately, 134 patients consented to participate. After excluding 5 patients due to late ineligibility, 129 patients were randomized.
Pre-assignment Details: A total of 188 eligible patients were approached for study participation. Of these, 54 declined for various reasons: not tech-savvy (n = 2), no time/too busy (n = 13), not interested in clinical research (n = 5), feeling overwhelmed (n = 10), other reasons (n = 6), and two or more of the aforementioned reasons (n = 18). Ultimately, 134 patients consented to participate. After excluding 5 patients due to late ineligibility, 129 patients were randomized.
Period: Overall Study
Arm/Group | Arm I (Telemonitoring) | Arm II (Enhanced Usual Care)
Started | 64 | 65
Completed | 55 | 59
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Telemonitoring) | Arm II (Enhanced Usual Care) | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [47 to 64] | 52 [48 to 65] | 53 [47 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 24 | 56
  Male | 32 | 41 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 20 | 33
  Not Hispanic or Latino | 51 | 45 | 96
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 11 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 31 | 41 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 64 | 65 | 129

OUTCOME MEASURES:

1. Primary Outcome: Patient Postoperative Complications Using the Comprehensive Complications Index (CCI)
Description: Postoperative complications occurring within 30 days post-discharge after cancer surgery were measured using the Comprehensive Complications index (CCI), a validated tool that aggregates the Clavien grades of postoperative complications on a continuous scale ranging from 0 (no complication) to 100 (death).
Time Frame: Outcomes are measured up to 30 days post-discharge after cancer surgery. Duration of hospitalization: Median, 5 days (Min: 0, Max: 18).
Population: Eight of the 129 randomized patients did not provide data for this outcome due to aborted surgery.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm I (Telemonitoring) | Arm II (Enhanced Usual Care)
Number analyzed (Participants) | 62 | 59
score on a scale | 0 [0 to 8.7] | 0 [0 to 8.7]

2. Primary Outcome: Number of Participants Who Completed >= 70% of the Study
Description: Study completion was assessed based on the percentage of patients who completed at least 70% of the following during the study period: (a) daily step counts, (b) quality of life measures, and (c) patient-generated health data. These measures were assessed from baseline through 30 days post-discharge after cancer surgery.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Telemonitoring) | Arm II (Enhanced Usual Care)
Number analyzed (Participants) | 64 | 65
Participants
  Daily step counts | 54 | 56
  Quality of life measures | 54 | 58
  Patient-generated health data | 54 | 57

3. Primary Outcome: Number of Participants Who Reported Intervention Acceptability
Description: Acceptability of telemonitoring was assessed using a patient satisfaction tool administered within 30 days post-discharge after cancer surgery. The tool evaluated ease of use, time burden of participation, and access to technology.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Telemonitoring) | Arm II (Enhanced Usual Care)
Number analyzed (Participants) | 64 | 65
Participants | 50 | 52

4. Secondary Outcome: Participant Reported Symptom Severity Score as Measured by the MD Anderson Symptom Inventory (MDASI)
Description: The MDASI assesses the severity of symptoms at their worst in the last 24 hours on a 0-10 scale, with 0 being "not present" and 10 being "as bad as you can imagine." Scores from baseline to 30 days post-discharge were calculated. A linear mixed effects model (adjusted for baseline scores) was used to assess differences in symptom severity between both arms over time.
Time Frame: Outcomes are measured at baseline, 2 days, 7 days, 14 days, and 30 days post-discharge.
Population: Due to attrition in the study, the number of patients assessed at baseline differs from the number of patients analyzed during follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm I (Telemonitoring) | Arm II (Enhanced Usual Care)
Number analyzed (Participants) | 64 | 65
score on a scale
  Baseline | 1.81 [1.5 to 2.1] | 1.73 [1.4 to 2.0]
  Day 2 post-discharge: number analyzed (Participants) | 53 | 53
  Day 2 post-discharge | 2.63 [2.3 to 3.0] | 2.92 [2.6 to 3.3]
  Day 7 post-discharge: number analyzed (Participants) | 51 | 55
  Day 7 post-discharge | 1.74 [1.4 to 2.1] | 2.27 [1.9 to 2.6]
  Day 14 post-discharge: number analyzed (Participants) | 48 | 55
  Day 14 post-discharge | 1.48 [1.11 to 1.8] | 2.2 [1.9 to 2.5]
  Day 30 post-discharge: number analyzed (Participants) | 50 | 54
  Day 30 post-discharge | 1.21 [0.9 to 1.6] | 2.05 [1.7 to 2.4]

5. Secondary Outcome: Participant Reported Quality of Life as Measured by the EQ-5D-5L.
Description: The EQ-5D-5L descriptive system of 5 health dimensions includes 5 response categories of no problem, slight problems, moderate problems, severe problems, and extreme problems. The 5 responses give a health state or profile represented by a 5-digit number (for example, 12231) corresponding to response categories reported by patients. Health states are scored to give the EQ-5D-5L index using a scoring algorithm from a value set derived from valuation tasks typically undertaken with general population samples. Index scores range from -0.59 to 1 where 1 is the best possible health state. Scores from baseline to 30 days post-discharge were calculated. A linear mixed effects model (adjusted for baseline scores) was used to assess differences in QoL scores between both arms over time.
Time Frame: Outcomes are measured at baseline, 2 days, 7 days, 14 days, and 30 days post-discharge.
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm I (Telemonitoring) | Arm II (Enhanced Usual Care)
Number analyzed (Participants) | 63 | 65
score on a scale
  Baseline | 0.86 [0.8 to 0.9] | 0.85 [0.8 to 0.9]
  Day 2 post-discharge: number analyzed (Participants) | 53 | 53
  Day 2 post-discharge | 0.57 [0.5 to 0.6] | 0.54 [0.5 to 0.6]
  Day 7 post-discharge: number analyzed (Participants) | 51 | 55
  Day 7 post-discharge | 0.69 [0.6 to 0.7] | 0.61 [0.6 to 0.7]
  Day 14 post-discharge: number analyzed (Participants) | 48 | 55
  Day 14 post-discharge | 0.72 [.07 to 0.8] | 0.67 [0.6 to 0.7]
  Day 30 post-discharge: number analyzed (Participants) | 50 | 54
  Day 30 post-discharge | 0.8 [0.7 to 0.9] | 0.75 [0.7 to 0.8]

6. Secondary Outcome: Number of Participants Utilizing Healthcare Resource Use (Hospital Readmission)
Description: Differences in the number of patients readmitted to the hospital for an overnight stay within 30 days post-discharge were compared between the two study arms using the Chi-square test or Fisher's exact test.
Time Frame: Up to day 30 post-discharge
Population: Eight of the 129 randomized patients did not provide data for this outcome due to aborted surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Telemonitoring) | Arm II (Enhanced Usual Care)
Number analyzed (Participants) | 62 | 59
Participants | 10 | 13

ADVERSE EVENTS:
Time Frame: This is an intervention trial lasting three months post-treatment, with no blood draws, procedures, or other invasive assessments. Since this is not a drug trial, patients were not monitored for specific adverse events. However, one patient died prior to study participation. Each participant was monitored for mortality during the three-month post-discharge period.
Description: Since this is not a drug trial, adverse events were not recorded.
Arm/Group | Arm I (Telemonitoring) | Arm II (Enhanced Usual Care)
All-Cause Mortality (participants affected / at risk) | 0/64 | 1/65
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT04986566/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT04986566/ICF_000.pdf